CLINICAL TRIAL: NCT02164721
Title: Multicenter Automatic Defibrillator Implantation Trial - Chemotherapy-Induced Cardiomyopathy
Acronym: MADIT-CHIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Valentina Kutyifa, Principal Investigator, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MADIT-CHIC
Record Dates: First submitted 2014-06-12; First posted 2014-06-17 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Cardiomyopathy
Keywords: Heart failure; Chemotherapy-induced cardiomyopathy; Cardiac resynchronization therapy
MeSH Terms: conditions — Cardiomyopathies; Heart Failure | interventions — Defibrillators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CRT-D (Defibrillator) (Other): Implantation of a three-lead CRT-D (Defibrillator) in all registered patients
  Interventions: Device: Three-lead CRT-D (Defibrillator)

INTERVENTIONS:
Device: Three-lead CRT-D (Defibrillator) — The three-lead CRT-D (Defibrillator) will consist of a pulse generator, a right atrial lead, a right ventricular lead and a left ventricular lead.

SUMMARY:
The purpose of this trial or study is to determine if cardiac resynchronization therapy (CRT) can be a benefit to people who have impaired heart function due to past treatment with chemotherapy and/or chest radiation. The investigators are looking to enroll approximately 30 eligible subjects with heart failure in this trial. All patients enrolled and registered in the study will be implanted with a cardiac resynchronization therapy device that includes an implantable cardiac defibrillator (CRT-D). Clinical histories, physical exams, and external device testing will be collected both at the time of enrollment in the trial and during follow-up study visits. Following implantation of the CRT-D, patients will be contacted by phone at 3 months and will have a scheduled clinic visit follow-up at 6 months.

DETAILED DESCRIPTION:
With the advent of new therapies and an increasing number of long-term cancer survivors, the incidence and consequently the interest in chemotherapy-induced cardiomyopathy (CHIC) have been increasing. CHIC is a dose-dependent cardiomyopathy and presents as congestive heart failure several months to years after the administration of chemotherapy and/or chest radiation that includes the heart.

Greater than one-half of the patients exposed to just this class of drugs will show evidence of cardiac dysfunction, with 5% presenting with overt symptomatic heart failure. The overall incidence of CHIC is significantly underestimated as within the US alone, greater than 60,000 patients receive just anthracyclines every year. Despite this, there is little data on their response to conventional heart failure therapy. There is some preliminary evidence from two small, retrospective case-series suggesting that patients with CHIC and evidence of conduction tissue disease (i.e. a wide electrocardiographic depolarization duration (QRS) may significantly benefit from cardiac resynchronization therapy (CRT).

MADIT-CHIC is a multicenter, non-randomized, prospective observational study. The primary aim is to determine if CRT-D (Defibrillator) in high-risk patients with chemotherapy-induced cardiomyopathy will significantly improve left ventricular ejection fraction (LVEF) by echocardiography within 6 months of initiating CRT without adversely affecting mortality.

The study will last 6 months and will be conducted in 10-15 clinical centers in the United States.

Following implantation of the CRT-D device (Defibrillator), patients will be followed for 6 months. The first follow-up contact will be by phone at which time study personnel will review the patient's health status. The last study contact will be a 6-month clinic visit. At the 6-month visit, the patient's health status will be reviewed, the functioning of the CRT-D (Defibrillator) will be tested and an echocardiogram will be conducted. After the 6-month visit, the study-required follow-up will have been completed and patients will continue to have CRT-D (Defibrillator) clinical follow-up based on their physicians direction.

During the course of the study, Subjects will as outlined in the inclusion criteria continue on stable optimal pharmacologic therapy for the cardiac condition that is guideline-based and may include one or more of the following medications: Loop diuretics, Angiotensin converting enzyme (ACE) inhibitors and/or angiotensin receptor blocker (ARB), Aldosterone antagonists and/or Beta-blockers unless the subject is not indicated, contraindicated, or is intolerant of medication.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 (or of legal age to give informed consent specific to state and national law) up to 80 years of age
* Male or Female
* Without clinical heart failure at initiation of chemotherapy/radiation-induced treatment for an underlying malignancy, but developed clinical heart failure (cardiomyopathy: reduced left ventricular ejection fraction (LVEF) with a left bundle branch block (LBBB)-type of conduction disturbance; see next inclusion item) 6 months or more after initiation of the chemotherapy without other evident cause of the cardiomyopathy.
* Eligible for implantation of a CRT-D (cardiac resynchronization therapy-defibrillator) device according to one of the following options in currently available guidelines:

  1. Class 1: Left ventricular ejection fraction (LVEF) less than or equal to 35% AND sinus rhythm AND LBBB (left bundle branch block) with a QRS (electrocardiographic depolarization duration) duration greater than or equal to 150ms AND NYHA (New York Heart Association) class II, III or ambulatory IV symptoms on guideline-directed medical therapy
  2. Class 2a1: Left ventricular ejection fraction (LVEF) less than or equal to 35% AND sinus rhythm AND left bundle branch block (LBBB) with a QRS (electrocardiographic depolarization duration) duration 120-149ms AND New York Heart Classification (NYHA) class II, III or ambulatory IV symptoms on guideline-directed medical therapy
  3. Class 2a2: Left ventricular ejection fraction (LVEF) less than or equal to 35% AND sinus rhythm AND Non-left bundle branch block (LBBB) with a QRS(electrocardiographic depolarization duration) duration greater than or equal to 150ms AND New York Heart Classification (NYHA) class III or ambulatory IV symptoms on guideline-directed medical therapy
* On stable optimal pharmacologic therapy for the cardiac condition that is guideline-based and may include one or more of the following medications: Loop diuretics, Angiotensin converting enzyme (ACE) inhibitors and/or angiotensin receptor blocker (ARB), Aldosterone antagonists and/or Beta-blockers unless the subject is not indicated, contraindicated, or is intolerant of medication.

Exclusion Criteria:

* Currently implanted pacemaker or implantable cardioverter defibrillator (ICD) device
* Previous implant with a CRT (cardiac resynchronization therapy)/CRT-D (cardiac resynchronization therapy-defibrillator) device
* Cardiac condition not presumed to be caused by chemotherapy
* Documented symptoms or hemodynamically unstable ventricular tachyarrhythmia
* On active chemotherapy (must be at least 6 calendar months after last chemotherapy)
* Permanent or chronic Atrial Fibrillation (AF), or cardioversion for AF within the past 3 calendar months before consent date
* Structural heart disease such as congenital heart disease, valvular heart disease, e.g., rheumatic valvular heart disease, amyloid heart disease, etc.
* Coronary artery bypass graft surgery or percutaneous coronary intervention within the past 3 calendar months before consent date
* Enzyme positive myocardial infarction within the past 3 calendar months prior to consent date
* Unstable angina requiring hospitalization, with diagnostic work up and intervention within the past 3 months prior to consent date
* Angiographic evidence of coronary disease who are candidates for coronary revascularization and are likely to undergo coronary artery bypass graft surgery or percutaneous coronary intervention in the foreseeable future
* Class IV and expected to undergo transplant within study duration
* Current or past history of drug addiction or abuse that caused cardiomyopathy
* Pregnant or plans to become pregnant during the course of the trial.
* Recent cerebral vascular accident or transient ischemia attack within the previous 3 months prior to consent date
* Presence of any disease, other than the subject's cardiac or cancer disease, associated with a reduced likelihood of survival for the duration of the trial, e.g., uremia, liver failure, active malignant disease, etc.
* Participating in any other clinical trial
* Unwilling or unable to cooperate with the protocol
* Lives at such a distance from the clinic that travel for follow-up visits would be unusually difficult
* Does not anticipate being a resident of the area for the scheduled duration of the trial
* Unwilling to sign the consent for participation
* Physician does not allow participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD, PhD, Principal Investigator — University of Rochester
Locations (9):
- United States (9):
  - UCLA Cardiovascular Center, Los Angeles, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - New York Presbyterian Hospita/Columbia University Medical Center, New York, New York
  - Univeristy of Rochester Medical Center, Rochester, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Singh JP, Solomon SD, Fradley MG, Barac A, Kremer KA, Beck CA, Brown MW, McNitt S, Schleede S, Zareba W, Goldenberg I, Kutyifa V; MADIT-CHIC Investigators. Association of Cardiac Resynchronization Therapy With Change in Left Ventricular Ejection Fraction in Patients With Chemotherapy-Induced Cardiomyopathy. JAMA. 2019 Nov 12;322(18):1799-1805. doi: 10.1001/jama.2019.16658. PMID 31714987

RESULTS

PARTICIPANT FLOW:
Groups:
- CRT-D (Defibrillator): Implantation of a three-lead Cardiac Resynchronization Therapy -Defibrillator (CRT-D) in all registered patients
  Three-lead CRT-D (Defibrillator): The three-lead CRT-D (Defibrillator) will consist of a pulse generator, a right atrial lead, a right ventricular lead and a left ventricular lead.
Period: Overall Study
Arm/Group | CRT-D (Defibrillator)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CRT-D (Defibrillator)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [54 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 21
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30
Number of participants with Nonischemic cardiomyopathy [Count of Participants; unit: Participants] — Population: In one patient, the presence of nonischemic cardiomyopathy was unknown.
  Participants
    number analyzed (Participants) | 29
    (all) | 29
Median Electrocardiographic depolarization duration (QRS) after consent [Median (Inter-Quartile Range); unit: ms] | 152 [142 to 160]
Number of participants with Left bundle branch block (LBBB) after consent [Count of Participants; unit: Participants] — Left Bundle Branch Block (LBBB) was ascertained by reviewing ECGs collected at baseline, following informed consent.
  Participants | 30
Sinus rhythm after consent [Count of Participants; unit: Participants] — Number of Participants with Normal Sinus Rhythm at Baseline.
  Normal Sinus Rhythm at Baseline was ascertained by reviewing ECGs collected at baseline, following informed consent.
  Participants | 29
Number of participants with Diabetes [Count of Participants; unit: Participants] | 6
Number of participants with Hypertension [Count of Participants; unit: Participants] | 17
Number of participants with a History of ventricular arrhythmias [Count of Participants; unit: Participants] | 3
Number of participants with a history of atrial arrhythmias [Count of Participants; unit: Participants] | 8
Number of participants with Anthracycline history [Count of Participants; unit: Participants] — Population: One patient had missing data for anthracycline history.
  Participants
    number analyzed (Participants) | 29
    (all) | 24
Median Time since cancer diagnosis [Median (Inter-Quartile Range); unit: years] | 13.8 [1.1 to 26.5]
Median Age at cancer diagnosis [Median (Inter-Quartile Range); unit: years] | 52 [40 to 59]
Number of participants with History of breast cancer [Count of Participants; unit: Participants] | 22
Number of participants with a History of leukemia or lymphoma [Count of Participants; unit: Participants] | 6
Number of participants with a History of sarcomas [Count of Participants; unit: Participants] | 2
Median blood urea nitrogen levels [Median (Inter-Quartile Range); unit: mg/dl] — Population: Data were available in 27 out of 30 participants.
  mg/dl
    number analyzed (Participants) | 27
    (all) | 20 [15 to 27]
Median Creatinine Levels [Median (Inter-Quartile Range); unit: mg/dl] — Population: Data were available in 28 out of 30 participants.
  mg/dl
    number analyzed (Participants) | 28
    (all) | 0.95 [0.85 to 1.25]
New York Heart Association class, II [Count of Participants; unit: Participants] — Heart failure symptom severity was categorized using the New York Heart Association (NYHA Class) at enrollment, stages below:
  I No limitation of physical activity. II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath.
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or shortness of breath.
  IV Unable to carry on any physical activity without discomfort with symptoms at rest.
  Participants | 17
New York Heart Association class, III [Count of Participants; unit: Participants] — Heart failure symptom severity was categorized using the New York Heart Association (NYHA Class) at enrollment, stages below:
  I No limitation of physical activity. II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath.
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or shortness of breath.
  IV Unable to carry on any physical activity without discomfort with symptoms at rest.
  Participants | 13
Median Blood pressure, systolic [Median (Inter-Quartile Range); unit: mm Hg] | 121.5 [116 to 133]
Median Blood pressure, diastolic [Median (Inter-Quartile Range); unit: mm Hg] | 70.5 [60 to 77]
Number of participant taking a Beta-Blocker [Count of Participants; unit: Participants] | 28
Angiotensin-Converting Enzyme Inhibitor (ACEI) or Angiotensin Receptor Blocker (ARB) [Count of Participants; unit: Participants] | 23
Number of participants taking a Loop diuretic [Count of Participants; unit: Participants] | 28
Number of participants taking Aldosterone [Count of Participants; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular Ejection Fraction
Description: The primary endpoint will be the change in left ventricular ejection fraction (LVEF) from baseline to six months
Time Frame: 6 months post implant
Population: Change in left ventricular ejection fraction (LVEF) from baseline to six months was analyzed with 26 patients with data available.
Measure: Mean (Standard Deviation); unit: percentage of LVEF
Arm/Group | CRT-D (Defibrillator)
Number analyzed (Participants) | 26
percentage of LVEF | 10.6 (6.6)

2. Secondary Outcome: Number of Participants With All-Cause Mortality
Description: Number of Participants with All-Cause Mortality in CRT-D patients
Time Frame: 6 months post implant
Population: Event rate of all-cause mortality is described.
Measure: Number; unit: participants
Arm/Group | CRT-D (Defibrillator)
Number analyzed (Participants) | 30
participants | 0

3. Secondary Outcome: Effects of CRT Therapy on Left Ventricular Volume at End Diastole
Description: Determine based on echocardiogram study if CRT therapy improves left ventricular volume at end diastole (LVEDV) between baseline and six months
Time Frame: 6 months post implant
Population: Describe 23 patients with data available on LVEDV change
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | CRT-D (Defibrillator)
Number analyzed (Participants) | 23
ml | -31.9 (22.5)

4. Secondary Outcome: Effects of CRT Therapy on Left Ventricular Volume at End Systole
Description: Determine based on echocardiogram study if CRT therapy improves left ventricular volume at end systole (LVESV) between baseline and six months
Time Frame: 6 months post implant
Population: Describe changes in LVESV in 23 patients with data available
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | CRT-D (Defibrillator)
Number analyzed (Participants) | 23
ml | -37.0 (20.4)

5. Other Pre Specified Outcome: Change in New York Heart Association (NYHA) Functional Class
Description: Improvement in NYHA functional class between baseline and six months (yes/no), ie. change from NYHA class III to NYHA II.
Time Frame: 6 months post implant
Population: Improvement in NYHA functional class between baseline and six months (yes/no) in 29 participants with data available.
Measure: Number; unit: participants
Arm/Group | CRT-D (Defibrillator)
Number analyzed (Participants) | 29
participants | 12

6. Other Pre Specified Outcome: Change in Left Atrial Size
Description: Change in left atrial size between baseline and six months
Time Frame: 6 months post implant
Population: Change in left atrial size between baseline and six months was analyzed in 26 patients with data available.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | CRT-D (Defibrillator)
Number analyzed (Participants) | 26
ml | -12.6 (9.6)

7. Other Pre Specified Outcome: Effects of CRT on Frequency of Heart Failure
Description: Effects of CRT on the frequency of heart failure with end point of inpatient hospitalization with augmented treatment for heart failure
Time Frame: 6 months post implant
Population: Frequency of heart failure described in the study population.
Measure: Number; unit: participants
Arm/Group | CRT-D (Defibrillator)
Number analyzed (Participants) | 30
participants | 1

ADVERSE EVENTS:
Time Frame: We have collected data on adverse events during the 6 months follow-up in the study.
Description: The definition of adverse event and/or serious adverse event is the same as on clinicaltrials.gov.
Arm/Group | CRT-D (Defibrillator)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 4/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-D (Defibrillator) (N=30)
Device Infection (Cardiac disorders) | 1 (1) — Device Pocket Infection (>30 days post-implant)
Pericardial effusion (Cardiac disorders) | 1 (1)
Inappropriate device therapy (Cardiac disorders) | 1 (1)
Shingles (Nervous system disorders) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) — Heart failure event with syncope related to heart failure, hypokalemia, and renal insufficiency
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-D (Defibrillator) (N=30)
Hypertension (Cardiac disorders) | 2 (2)
Atrial fibrillation/flutter (Cardiac disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The findings are limited by the small sample size, short follow-up, and absence of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT02164721/Prot_SAP_000.pdf